CLINICAL TRIAL: NCT06786975
Title: EFFECTIVENESS, ACCEPTABILITY AND ORAL HEALTH-RELATED QUALITY OF LIFE OF SILVER DIAMINE FLUORIDE COMPARED TO ATRAUMATIC RESTORATIVE TREATMENT FOR THE MANAGEMENT OF EARLY CHILDHOOD CARIES: PROTOCOL OF A PRAGMATIC RANDOMIZED CLINICAL TRIAL
Brief Title: Effectiveness and Acceptability of SDF Compared to ART for the Management of Early Childhood Caries
Acronym: SDF and ART
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de La Frontera (Other)
Responsible Party: Principal Investigator, Patricia Muñoz Millán, Public Health Master, Specialist in Paediatric Dentistry, PhD exam passed at the Universidad Autónoma de Barcelona, Universidad de La Frontera
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DI19-0091
Record Dates: First submitted 2024-12-05; First posted 2025-01-22 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Early Childhood Caries; Health Care Acceptability
Keywords: Early Childhood Caries; Silver Diamine Fluoride; Atraumatic Restorative Treatment
MeSH Terms: conditions — Patient Acceptance of Health Care | interventions — Dental Atraumatic Restorative Treatment

STUDY DESIGN:
Intervention Model Description: An open-label parallel superiority randomized clinical trial (RCT)
  Participants will be children with informed consent previously by their parents/guardians and assent given by the child. The participants will be randomized into two groups/arms with the permuted block randomization method, assuming an average of 3 teeth with caries lesions per child:
  * Experimental: 78 participants (children) for silver diamine fluoride application.
  * Control: 78 participants (children) for atraumatic restorative treatment technique.
  It's expected to have at least 234 teeth with caries lesions per group and 468 teeth with caries lesions in total. The child will be assigned as the unit of randomization, so all they teeth will be treated with the same intervention.
  Controls will be done up to 18 months after treatment (at 6, 12 and 18 months).
Masking Description: Considering the treatment types, it is not possible to mask operators, examiners or participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Silver Diamine Fluoride (Experimental): Participants who will receive oral health education and Silver Diamine Fluoride application in decayed teeth every 6 month. Controls will be made up to eighteen months.
  Interventions: Device: Silver Diamine Fluoride
- Atraumatic Restorative Treatment (Active Comparator): Participants who will receive oral health education and atraumatic restorative treatment in decayed teeth. Controls will be made every 6 months up to eighteen months, in case of restoration failure it will be made again.
  Interventions: Procedure: Atraumatic Restorative Treatment

INTERVENTIONS:
Device: Silver Diamine Fluoride — Tooth will be isolated with cotton rolls, the oral cavity will be dried with small cotton balls and the gingiva around the tooth, and surrounding structures, will be protected with vaseline. Then the silver diamine fluoride solution will be applied to cavitated caries lesions with a micro applicator for one minute approximately. If necessary the solution excess should be removed with a gauze.
  Finally the child's teacher will be given the indications for the child to not eat, drink or rinse up to 30 minutes after the treatment, and to evaluate if any sign or symptom related to the tooth appears.
  Other Names: Silver dental arrest; Diammine silver fluoride dental hypersensitivity varnish
  Arms: Silver Diamine Fluoride
Procedure: Atraumatic Restorative Treatment — Participants will be treated with Atraumatic Restorative Treatment (ART) technique. Glass ionomer will be used for cavity filling (Ketac MolarTM, 3M ESPETM) according to manufacter specifications and will be applied with a spatula, followed by finger pressure using vaseline for a few seconds; for occluso-proximal cavities, a matrix band will be used. The restoration will be protected with vaseline and then the occlusion will be checked with articular paper after the initial adjustment (approximately 5 minutes). Finally the child's teacher will be given the indications for the child to not eat, drink or rinse up to 30 minutes after the treatment, and to evaluate if any sign or symptom related to the tooth appears.
  Arms: Atraumatic Restorative Treatment

SUMMARY:
The goal of this clinical trial is to assess the acceptability and clinical effectiveness of Silver Diamine Fluoride (SDF) in comparison with Atraumatic Restorative Treatment (ART) in Early Childhood Caries (ECC) management at the community level. The main question it aims to answer are:

• It's SDF more accepted and effective than ART in early childhood caries management when implemented at the community level?

Participants will be diagnosed by an experienced and calibrated dentist using the International Caries Detection and Assessment System (ICDAS), then children with decayed teeth will be treated with SDF (experimental) or ART (control); another operator will choose randomly the treatment for each participant. Furthermore, oral health education component will be given to children, parents and educators.

Follow-up visits will be made at 6 and 12 months after child's treatment is complete. Before and after treatment parents will be asked to complete a child personal background survey (before), Early Childhood Oral Health Impact Scale (ECOHIS) questionnaire (before and at follow-ups) and a oral health satisfaction survey (one week after treatment and at follow-ups). The acceptability will be assessed through quantitative and qualitative methods.

Researchers will compare the SDF's groups and the ART's group to see which of them is more accepted and effective.

DETAILED DESCRIPTION:
An open-label parallel superiority randomized clinical trial (RCT) will be conducted involving children aged 2 to 5 years.

The aim of this clinical trial is to assess the acceptability and clinical effectiveness of Silver Diamine Fluoride (SDF) in comparison with Atraumatic Restorative Treatment (ART) in Early Childhood Caries (ECC) management. As well, this clinical trial sought to compare the oral health quality of life related and to contrast possible adverse effects between both therapies.

Participants will be screened and diagnosed by an experienced and calibrated dentist using the International Caries Detection and Assessment System (ICDAS), thereafter only children with decayed teeth (or tooth) will be treated. After the diagnostic participants eligibles will be randomly chosen by another operator to be treated with SDF or ART for all teeth who need treatment in the child:

* Experimental: SDF application in decayed teeth and oral health education component.
* Control: ART technique in decayed teeth and oral health education component.

The oral health education component will be given to children, parents and educators.

The eligible children parents will be asked to fulfill a children personal background survey (before treatment), the Early childhood oral health impact scale (ECOHIS) questionnaire (before and after treatment at follow-ups) and a oral health satisfaction survey (a week after treatment and at follow-ups). The acceptability will be assessed through quantitative and qualitative methods.

A sample is: 234 teeth with carious lesions per group is estimated. Estimating an average of three teeth with carious lesions per child, 78 children are necessary per group.

ELIGIBILITY:
Inclusion Criteria:

* Children belonging to INTEGRA or JUNJI kindergarten, from 2 years up to 5 years and 11 months with informed consent signed by parents and assent from the child.
* Children with at least one active cavitated caries lesion, extended in dentin with no signs of pulp involvement and diagnosed with ICDAS code 5.

Exclusion Criteria:

* Children with underlying systemic disease or disability
* Children with known allergies to dental materials used
* Children with transitory residence
* Children with severe alterations of the dental estructure

Ages: 24 Months to 71 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 156 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Arrest of the carious lesion: | 6 and 12 months
  The activity and inactivity of the lesion shall be assessed. A value of 0 shall be recorded if the lesion is inactive and a value of 1 if the lesion is active. For the assessment of activity, the parameters described in the Caries Care Guide shall be considered.
  For the Fluoride Diamine Silver group, the lesion's surface should have a shiny appearance and hard consistency on examination to be considered inactive, when a soft, leathery and plaque retentive tissue is present, the lesion shall be considered active. For the Atraumatic Restorative Technique group, the Caries Associated to Restoration or Sealant (CARS)* criteria will be applied, being considered inactive if the margin is intact (good margin) and upon presentation of a restoration or plaque retentive sealant requiring adjustment or replacement will be considered active.
  [*CARS includes 3 categories: good margin; defective (plaque-retentive, can be adapted); defective(needs replacement)]
Parental acceptability: quantitative measure | 1 month, 6 months, and 12 months
  Parental acceptability will be measured through a survey at 1 month, 6 months, and 12 months post-treatment following by a own elaboration questionnare.The survey includes 6 questions. Whether they would recommend the treatment based on the results (aesthetics, absence of pain, arrest of lesion) and experience of the treatment received by their child (adaptation and access to care).
Parental acceptability: qualitative measure | 1 month
  A qualitative method will be used through semi-structured interviews to be conducted one month after the intervention.Parents with the lowest (10th percentile) and highest (90th percentile) acceptability (Parental acceptability: quantitative measure) will be selected. The semi-structured interview will explore their child's experience, what factors lead them to feel satisfied/dissatisfied with the treatment, factors that influenced their child's perceived comfort or discomfort during treatment, relevance of aesthetics, importance of the care setting to their satisfaction or dissatisfaction.
Children's acceptability | at the end of the initial treatment, 6 and 12 months.
  Children's acceptability of treatment as assessed by the operator using Frankl´s scale at the end of the initial treatment, 6 and 12 months. The minimum value=1 and the maximum value is 4. The higher scores mean a worse children's acceptability. [Frankl´s scale was used to evaluate child's behavior in the dental setting in four categories: 1-definitely negative 2-negative 3-positive 4- definitely positive]
Change in oral health-related quality of life (OHRQoL) | baseline and 6 months
  Description: Change in oral health-related quality of life will be measured by the difference in the ECOHIS score between baseline and 6 months. The ECOHIS is a proxy-reported questionnaire for measuring the OHRQoL of preschool children and their families. It comprises of 13 items, covering six domains in two sections. The child's impacts section contains 4 domains. The family's impacts section contains 2 domains. Response categories for each question are rated on a 5-point Likert scale to record how often an event has occurred during the child's life: 0 = never, 1 = hardly ever, 2 = occasionally, 3 = often, 4 = very often, and 5 = don't know. ECOHIS scores are calculated as a simple sum of the response codes for the child and family sections separately and also a total score. The minimum value is 0 and maximum value is 52. Higher scores mean a worse quality of life.

SECONDARY OUTCOMES:
Absence of pulp pathology | 6 and 12 months
  Absence of pulp pathology: pufa=0 Measured with pufa index* [*pufa= 1 o >1 If presents p: pulpal involvement, opening of pulp chamber is visible or coronal tooth structures are destroyed by caries u: ulceration, traumatic ulceration in the soft tissues (tongue and mucosa), caused by tooth or root fragments f: a sinus tract releasing pus originating from an abscess and opening into the oral cavity a: abscess, dento-alveolar abscess.]
Presence of the tooth in the mouth. | 6 and 12 months
  Presence of the tooth in the mouth. This refers to the fact that the tooth that was treated is still present in the mouth at the time of the control examination and has not been surgically extracted. It will be valued as 0 if it is present and as 1 if it has been extracted.
Presence of adverse effects | 6 and 12 months
  A questionnaire will be applied to the parents a week after treatment and also at 6 and 12 months follow-ups after treatment, where they'll have to report the presence of any adverse effect related to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Muñoz, Master, Study Director — Universidad de La Frontera; Patricia Pineda, Master, Study Chair — Universidad de La Frontera; Carlos Zaror, Doctor, Study Chair — Universidad de La Frontera
Locations (1):
- Universidad de La Frontera, Temuco, La Araucanía, Chile

IPD SHARING:
Plan to Share IPD: Yes
Data sharing plan:
  Study Protocol, Statistical Analysis Plan, Informed Consent Form will be available in the published protocol. The final, anonymized individual participant data (including the statistical code) that underlie the results will be available upon reasonable request. Data sharing will commence after the publication of the primary results and remain accessible for a minimum of five years. Proposals must be methodologically sound and sent to patricia.munoz@ufrontera.cl. Data users must formally sign a Data Access Agreement to ensure compliance with ethical guidelines and participant privacy. Shared data will strictly exclude any direct or indirect identifiers. All researchers using the data must agree to acknowledge the original researchers and the trial's funding source.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Study protocol, statistical analysis plan, informed consent form will be available since February 2026. Analytic code will be available since January 2027
Access Criteria: The Data sharing Proposals must be methodologically sound and sent to patricia.munoz@ufrontera.cl. Data users must formally sign a Data Access Agreement to ensure compliance with ethical guidelines and participant privacy.